CLINICAL TRIAL: NCT07223034
Title: LU-TARGET: A Phase 1 Study of Lutetium-177-PSMA-617 Adjuvant Radiotherapy for IDH Wild Type Gliomas Expressing PSMA Following Standard Treatment
Brief Title: A Study of 177Lu-PSMA-617 in People With Gliomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-169
Record Dates: First submitted 2025-10-28; First posted 2025-10-31 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Glioma; Diffuse Astrocytoma, IDH-Wildtype (Grade 2-4); Glioblastoma, IDH-wildtype; Diffuse Midline Glioma, H3 K27-Altered; Diffuse Hemispheric Glioma, H3 G34-mutant; Diffuse Pediatric-type High-grade Glioma, H3-wildtype and IDH-wildtype
MeSH Terms: conditions — Glioma; Astrocytoma; Glioblastoma | interventions — Temozolomide; Pluvicto; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA-617 (Experimental): Patients will begin the first and second cycles of adjuvant Temozolomide (TMZ) the night before the first and second infusions of 177Lu-PSMA-617, respectively. Post-treatment, MRI of the brain will be obtained every 2 months, as per standard of care. A 68Ga-PSMA-PET scan will be performed with the MRI of the brain 1 month after the second cycle of 177Lu-PSMA-617 and again at evidence of disease progression.
  Interventions: Drug: Temozolomide; Drug: 177Lu-PSMA-617; Diagnostic Test: 68Ga-PSMA-PET scan/ MRI; Behavioral: Quality of Life Questionnaires

INTERVENTIONS:
Drug: Temozolomide — Patients will begin taking Temozolomide orally on the first 5 days of each 28-day cycle. The first dose will be given the evening before the first infusion of 177Lu-PSMA- 617.
Drug: 177Lu-PSMA-617 — This agent will be given for 2-6 total doses, spaced 4 weeks (+/-1 week) apart. This will be administered on the 2nd day of the first two cycles of SOC adjuvant temozolomide.
Diagnostic Test: 68Ga-PSMA-PET scan/ MRI — Approximately 4 weeks after cycle 2 of radiopharmaceutical therapy (RPT), patients will undergo post-treatment imaging with 68Ga- PSMA PET and MRI
Behavioral: Quality of Life Questionnaires — baseline assessments, QOL surveys will be conducted with XeQOL and FACT-Br at 6 months and 12 months post treatment

SUMMARY:
The researchers are doing this study to find out whether the radiopharmaceutical therapy (RPT) 177Lu-PSMA-617 is a safe treatment for people with IDH wild type glioma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed histologic diagnosis of a WHO grade 2-4 glioma that is IDH1 R132H-wildtype, including the following:

  * Diffuse astrocytoma, IDH-wildtype (grade 2-4)
  * Glioblastoma, IDH-wildtype
  * Diffuse midline glioma, H3 K27-altered
  * Diffuse hemispheric glioma, H3 G34-mutant
  * Diffuse pediatric-type high-grade glioma, H3-wildtype and IDH-wildtype PSMA positive pathological stain (by immunohistochemistry) of baseline (pre-radiotherapy) resection or biopsy sample
* Completion of standard of care therapy including surgery (for resectable tumors) and adjuvant EBRT for glioma
* Patients must be on a dose of 4 mg or less of dexamethasone (or dexamethasone equivalent steroid) for 5 days prior to first planned dose of radiopharmaceutical
* Age ≥ 18
* ECOG ≤ 2
* Serum creatinine level < 1.5 x ULN or EGFR > 60 mL/min
* Liver laboratory values: ALT and AST ≤ 2.5 x ULN; Albumin > 2 g/ dL; Bilirubin < 3 X ULN
* Normal organ and marrow function as defined as the following

  * Total white blood count > 3.0 K/mcL
  * ANC ≥ 1.5 K/mcL
  * Platelets ≥ 100 K/mcL
  * Hemoglobin ≥ 9 g/dL
* Adequate contraception prior to registration (see section 9.0)
* Ability to understand, and willingness to sign the informed consent.

Exclusion Criteria:

* Patient known to harbor any other non-canonical IDH mutations (i.e., non-R132H)
* Target lesion within 5 mm of either the brainstem, optic chiasm or optic nerves Receipt of bevacizumab as part of the initial treatment for glioma
* Life expectancy less than 12 weeks
* Nonhealing wound, ulcer or bone fracture
* History of severe brain injury
* Patient not eligible for sequential MRI evaluations
* Patients with prior RT to > 25% of the skeleton or prior exposure to prior Radium223, Strontium89 or Samarium153 containing compounds
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen
* Patients with known or suspected history of grade II or higher chronic kidney disease (CKD)
* Unable to tolerate the PSMA PET/MR or PSMA PET/CT
* History of viral hepatitis or chronic liver disease with active symptoms
* History of pituitary or adrenal dysfunction
* Previously diagnosed active infection (e.g., human immunodeficiency virus [HIV] or viral hepatitis)
* Any condition that in the opinion of the investigator, would preclude participation in this study
* Receipt of any other investigational agents or participation in a concurrent treatment protocol
* Known allergies, hypersensitivities, or intolerance to 68Ga-PSMA-11/177Lu-PSMA-617 or its inactive compounding components
* Current or planned pregnancy
* Refusal to comply with detailed contraception requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Descriptively report the toxicity | up to 8 weeks post first infusion
  using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  PFS will be defined as the time from treatment initiation to progression of disease as noted radiographically per RANO 2.0 criteria or death, whichever occurred first, and will be analyzed using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Imber, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/